CLINICAL TRIAL: NCT00805493
Title: Double-Blind Placebo-Controlled Trial of Riluzole in Pediatric Bipolar Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment of participants
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 090042; 09-M-0042 (Other: The National Institutes of Mental Health)
Record Dates: First submitted 2008-12-06; First posted 2008-12-09 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Bipolar Disorder; Anxiety Disorders; Bipolar Affective Disorder; Bipolar Depression
Keywords: Mania; Bipolar; Bipolar Disorder; Bipolar Manic-Depressive Illness; Bipolar Mood Disorder
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders; Mania | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication Taper (No Intervention): All participants begin with gradual tapering to the point of discontinuing medication
- Random assignment to placebo (No Intervention): Once they are medication-free, 50% of participants are randomized to placebo
- Random assignment to riluzole (Active Comparator): One they are medication-free, 50% of participants are randomized to riluzole
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole
  Arms: Random assignment to riluzole

SUMMARY:
Pediatric Bipolar Disorder (BD) is uncommon in children. Its symptoms include periods of manic behavior (being overly happy or giddy, feeling grandiose, feeling a decreased need for sleep, having too much energy, moving more than usual, talking fast, having speeded-up thoughts and other symptoms). Sometimes there also is depression (extreme feelings of sadness or irritability, not taking pleasure in things, even ones that used to be enjoyable, feeling worthless or guilty, sleeping too much or having trouble getting to or staying asleep, feeling slowed down or restless, having wishes to be dead or suicidal ideas, and other symptoms). Pediatric BD is often difficult to treat; children may respond only partially to the medications now available or have too many side effects to tolerate them.

Riluzole is a medication that is thought to work on a brain chemical called glutamate that may be involved in symptoms of depression and BD. Previous research studies have shown that riluzole may help adults with BD who have depression and adults who have depression, anxiety disorders, or obsessive-compulsive disorders. Riluzole may also be helpful for children with obsessive-compulsive disorder. However, it has never been given to children with BD.

This study will evaluate the effectiveness of riluzole in 80 patients between 9 and 17 years of age who have BD and symptoms of anxiety. Participants must have tried at least two other medications that have not been effective.

The study will consist of four phases carried out over 4 to 5 months. Most children will be inpatients at the Pediatric Behavioral Health Unit for at least part of the study.

In Phase 1, each patient will undergo blood and urine tests, and will gradually taper off his or her medication. The duration of this phase depends on the medication that the patient was receiving before starting the study.

In Phase 2, the patient will remain off all medication for 1 week. Throughout this time, patients will be monitored carefully and medication will be restarted if needed.

In Phase 3, which lasts 8 weeks, patients will be assigned randomly to receive only riluzole or only a placebo. Those who receive riluzole will have the dose adjusted as needed. Patients and families will be informed of which drug they were on at the end of this phase. Patients who improved on riluzole may continue to receive it from NIH for 1 month and will then be prepared for discharge from the study. Patients who received placebo and improved, and those who received riluzole but did not improve, will be treated with standard medications as appropriate and prepared for discharge from the study.

Phase 4 is for patients who received placebo and did not improve. They will be given the chance to try riluzole for 8 weeks and, if it is effective, continue it for an additional 4 weeks while they prepare to be discharged from the study.

Patients will not be able to receive riluzole at the National Institutes of Health after the completion of the study. However, the child's doctor may be able to prescribe riluzole as an off-label use.

Most patients will be admitted to the Pediatric Behavioral Health Unit at the National Institutes of Health Clinical Center during the medication withdrawal part of the study (Phases 1 and 2). From Phase 3 on, a patient may participate as an inpatient, outpatient, or in day treatment, depending on what is in his or her best interests.

All participants in this study will be invited to also enroll in the National Institute of Mental Health protocol 00-M-0198, The Phenomenology and Neurophysiology of Affective Dysregulation In Children And Adolescents With Bipolar Disorder. Some research tests for that protocol will be done during the medication-free period of this protocol.

...

DETAILED DESCRIPTION:
OBJECTIVE: To test the efficacy of riluzole in youth with bipolar disorder

STUDY POPULATION: Youth, ages 9-17, with DSM-IV bipolar disorder, who have failed to respond to two adequate trials of medication, one with an atypical antipsychotic medication, and the second with either a mood stabilizing medication or a second atypical antipsychotic medication.

DESIGN: Medication withdrawal, followed by a 15-day dose stabilization phase and a 6-week double-blind, placebo-controlled treatment trial. The first two phases will be completed as inpatients or in day treatment, while the third phase can be completed either in those settings or as an outpatient. Individuals who received placebo will be offered an 8-week open trial of riluzole followed by an additional 4 weeks if they respond, while those who received riluzole in the placebo-controlled trial and wish to continue it will receive 4 weeks of open treatment. Thus, all patients will have the opportunity to receive a total of 12 weeks of riluzole treatment.

OUTCOME MEASURES: Clinical rating scales, including the Pediatric Anxiety Rating Scale and the Clinical Global Improvement Scale

ELIGIBILITY:
* INCLUSION CRITERIA:
* Boys and girls
* Ages 9-17 years of age
* Meet DSM-IV criteria for bipolar disorder.
* The child must have a primary caregiver who can accompany him or her on trips to NIMH, provide reliable history and information, and complete rating scales.
* Patients must have a psychiatrist who provides clinical care for their BPD.
* All youth accepted into the study must be able to complete self-rating forms and to cooperate with other study procedures.
* Previous treatment failure as defined by:

  1. Failure to respond to an adequate trial (adequate dose for at least two weeks) of a mood stabilizer (either lithium or divalproex) plus an adequate trial (sufficient dose for an adequate duration) of an atypical antipsychotic (such as risperidone, olanzapine, quetiapine, ziprasidone, or aripiprazole)
  2. Failure to respond to an adequate trial (sufficient dose for an adequate duration) of two atypical antipsychotics (such as risperidone, olanzapine, quetiapine, ziprasidone, or aripiprazole) or
  3. Evidence of intolerance (severe weight gain or other side effects) of a mood stabilizer or atypical antipsychotic agent.
* The child is failing his/her current treatment as defined by (all 3 met):

  1. The child's current CGAS score must be less than 60.
  2. The child's current psychiatrist must agree that the child's response to his/her current treatment is no more than minimal or there are drug side effects that are proving problematic. According to this criterion, it would be clinically appropriate to change the child's current treatment.
  3. On the basis of record review and interviews with child and parent, the research team agrees that the child's response to his/her current treatment is no more than minimal.
* Subject has a PARS score of greater than or equal to 10, derived from the total of the following individual items: 3 (overall severity of anxious feelings), 5 (overall avoidance), 6 (interference with family), and 7 (interference outside of the home). In addition, patients must score 3 or higher (i.e., in the clinical range) on at least one of the four items noted above.

EXCLUSION CRITERIA:

* I.Q. less than 70
* Autistic disorder or severe pervasive developmental disorder; psychosis that interferes with the child's capacity to understand and comply with study procedures;
* Unstable medical illness (e.g. severe asthma) or contraindication to riluzole
* Medical illness that could cause the symptoms of bipolar illness (e.g. multiple sclerosis, thyroid disease);
* Pregnancy
* Renal or hepatic dysfunction that would interfere with excretion or metabolism of riluzole as evidenced by increase above upper limits of normal for BUN/creatinine, or two-fold elevation of serum transaminases (ALT/SGPT, AST/SGOT), gamma glutamate (GGT), or bilirubin.
* Documented history of hypersensitivity or intolerance to riluzole.
* Substance abuse within two months of study entry

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Leibenluft, MD, Principal Investigator — NIH, NIMH-IRP
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amiel JM, Mathew SJ. Glutamate and anxiety disorders. Curr Psychiatry Rep. 2007 Aug;9(4):278-83. doi: 10.1007/s11920-007-0033-7. PMID 17880858
- [Background] Axelson D, Birmaher B, Strober M, Gill MK, Valeri S, Chiappetta L, Ryan N, Leonard H, Hunt J, Iyengar S, Bridge J, Keller M. Phenomenology of children and adolescents with bipolar spectrum disorders. Arch Gen Psychiatry. 2006 Oct;63(10):1139-48. doi: 10.1001/archpsyc.63.10.1139. PMID 17015816
- [Background] Bensimon G, Lacomblez L, Meininger V. A controlled trial of riluzole in amyotrophic lateral sclerosis. ALS/Riluzole Study Group. N Engl J Med. 1994 Mar 3;330(9):585-91. doi: 10.1056/NEJM199403033300901. PMID 8302340

RESULTS

PARTICIPANT FLOW:
Groups:
- Riluzole: Those randomized to riluzole
- Placebo: Those randomized to receive placebo
- Not Randomized: Those who withdrew prior to the decision to randomize
Period: Overall Study
Arm/Group | Riluzole | Placebo | Not Randomized
Started | 3 | 2 | 1
Completed | 1 | 2 | 0
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Not Randomized | Total
Number analyzed (Participants) | 3 | 2 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 3 | 2 | 1 | 6
  BTWN | 0 | 0 | 0 | 0
  GTE65 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 1 | 2 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Hawaiian | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression--Improvement
Description: This is a clinician rated measure that is a standard in pharmacological trials. the scores range from 1 to 8 with 5 being unchanged, 1 being completely recovered and 8 being markedly worse.
Time Frame: 8 week trial with the study running for about 4 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Riluzole: The group randomized to riluzole
Arm/Group | Riluzole | Placebo | Not Randomized
Number analyzed (Participants) | 3 | 2 | 0
units on a scale | 4 (.82) | 4 (1) |

2. Primary Outcome: Pediatric Anxiety Scale
Description: A standard measure of severity of anxiety over the previous week. The score ranges from a total of 0-25, with 0 being absence of symptoms and impairment, and 25 being marked symptoms and severe impairment. The outcome measure for each participant is the change in PARS, that is, the difference at week 8 compared to baseline (when medication-free).
Time Frame: Weekly for 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: The group randomized to receive placebo
- Not Randomized: Participants who withdrew prior to the decision to randomize
- Riluzole: The group randomized to receive riluzole
Arm/Group | Placebo | Not Randomized | Riluzole
Number analyzed (Participants) | 2 | 0 | 3
units on a scale | 1.67 (3.09) |  | -2.5 (0.5)

ADVERSE EVENTS:
Arm/Group | Riluzole | Placebo | Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=3) | Placebo (N=2) | Not Randomized (N=1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations in enrollment led to early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes